CLINICAL TRIAL: NCT01722045
Title: An Open-Label Study of the Efficacy, Safety, and Tolerability of Intravitreal Administration of VEGF Trap-Eye (Intravitreal Aflibercept Injection) in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Study to Assess Best Corrected Visual Acuity (BCVA) in Patients With Neovascular Age-Related Macular Degeneration (AMD) Who Are Administered VEGF Trap-Eye (Intravitreal Aflibercept Injection)
Acronym: RE-VIEW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-AMD-1124
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Age - Related Macular Degeneration (AMD)
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label IAI (Experimental)
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection (IAI)

SUMMARY:
This is a phase 4, open-label, single arm, multicenter, clinical study in patients with neovascular AMD designed to evaluate the efficacy and safety of Intravitreal Aflibercept Injection (IAI) administered over 2 years , and to provide clinical information from the first year in the trial evaluating the adverse effects, if any, on the corneal endothelium following administration of IAI.

ELIGIBILITY:
Inclusion criteria include but are not limited to:

1. Men or women great than or equal to 50 years of age with unilateral neovascular AMD
2. BCVA ETDRS letter score of 73 to 24 (20/40 to 20/320) in the study eye
3. Active primary subfoveal choroidal neovascularization (CNV) lesions secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by FA in the study eye
4. The CNV area must be at least 50% of total lesion size
5. Willing and able to comply with clinic visits and study-related procedures
6. Provide signed informed consent
7. Provide signed Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion criteria include but are not limited to:

1. Neovascular AMD in the fellow eye
2. Corneal endothelial measures as judged by an independent reading center
3. Any prior use of intraocular anti-VEGF treatment for neovascular AMD in either eye
4. Structural damage to the center of the macula in the study eye that is likely to preclude improvement in BCVA following the resolution of macular edema
5. History of cataract surgery, or other intraocular surgery in either eye, within 1 year of screening
6. History of cataract surgery, or other intraocular surgery in either eye, within 1 year of screening, or yttrium aluminum garnet (YAG) Capsulotomy within 3 months of screening
7. Contact lens wear in either eye within 6 months of screening
8. History of angle closure glaucoma in either eye
9. Intraocular laser therapy including selective laser trabeculoplasty (SLT), YAG, prophylactic peripheral iridotomy (PI) in either eye within 1 year of screening, or YAG Capsulotomy within 3 months of screening
10. History of cataract surgery requiring an anterior chamber intraocular lens implant at any time in either eye
11. Any prior ocular trauma (blunt or penetrating) in either eye
12. Embedded corneal foreign body in either eye
13. Evidence of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye
14. Ocular media of insufficient quality to obtain fundus and OCT images in the study eye
15. Any prior ocular inflammation/infection in either eye within 3 months of the screening visit
16. Any prior use of amantadine
17. Significant pre-retinal fibrosis involving the macula in the study eye (where, in the opinion of the investigator, the pre-retinal fibrosis is causing distortion or traction on the central macular region which may be limiting vision, or inducing retinal edema/thickening, beyond that due to underlying CNV)
18. Intraocular pressure (IOP) greater than or equal to 30 mm Hg in the study eye at screening
19. Uncontrolled diabetes mellitus (DM) (HbA1c ≥8)
20. Current treatment with systemic anti-VEGF therapeutics at screening
21. Known serious allergy to the fluorescein sodium for injection in angiography
22. Participation in an investigational study within 30 days prior to the screening visit that involved treatment with any drug (excluding vitamins and minerals) or device.
23. Positive serum hCG pregnancy test at the screening visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (49):
- United States (49):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Oakland, California
  - Palm Desert, California
  - Sacramento, California
  - Santa Ana, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Pensacola, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Oak Park, Illinois
  - New Albany, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Jackson, Michigan
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Portsmouth, New Hampshire
  - Bloomfield, New Jersey
  - Lawrenceville, New Jersey
  - Northfield, New Jersey
  - Teaneck, New Jersey
  - Rochester, New York
  - Asheville, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Salem, Oregon
  - Kingston, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Florence, South Carolina
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Arlington, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 43 sites in the US from 14Nov2012 to 03Sep2015. The target study population consisted of men and women 50 years of age and older with neovascular AMD who met all study eligibility criteria. A total of 288 patients were screened, of whom 154 patients were enrolled and treated. A total of 126 patients completed week 100.
Groups:
- Open Label IAI: 2 mg IAI (Intravitreal Aflibercept Injection) at 4-week intervals (2Q4) up to week 8 for a total of 3 injections, and 2 mg at 8-week intervals (2Q8) thereafter until week 96
Period: Overall Study
Arm/Group | Open Label IAI
Started | 154
Completed | 126
Not Completed | 28
Not completed — Adverse Event | 8
Not completed — Death | 3
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 4
Not completed — Protocol Deviation | 1
Not completed — Physician Decision | 3
Not completed — Relocation (did not wish to transfer) | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was based on the safety analysis set (SAF) and included all patients who received at least 1 dose of study drug, regardless of the treatment for the study eye or the fellow eye.
Groups:
- Open Label IAI: Intravitreal Aflibercept Injection (IAI)
Arm/Group | Open Label IAI
Number analyzed (Participants) | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 137
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 58
Best Corrected Visual Acuity (BCVA) in the study eye (Letters Read) [Mean (Standard Deviation); unit: letters correctly read] — Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision.
  letters correctly read | 54.3 (13.47)
Central Subfield Thickness in the study eye by Optical Coherence Tomography (OCT) [Mean (Standard Deviation); unit: micrometers (μm)] — Retinal and lesion characteristics (wet or dry) were evaluated using spectral domain OCT on the study eye and the fellow eye at every study visit.
  micrometers (μm) | 420.5 (134.90)
Corneal Endothelial Cell Density - Endothelial Cell Density Evaluable Set (EES) [Mean (Standard Deviation); unit: cells/mm^2] — Central ECD of the corneal endothelium in the study eye and the fellow eye was evaluated by specular microscopy. Population: EES
  cells/mm^2
    Study eye: number analyzed (Participants) | 118
    Study eye | 2409.8 (363.89)
    Fellow eye: number analyzed (Participants) | 118
    Fellow eye | 2388.0 (383.93)

OUTCOME MEASURES:

1. Primary Outcome: Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score From Baseline to Week 100 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision. LOCF approach was used if any ETDRS letter score was missed after start of treatment, but baseline data were not carried forward. No formal statistical analyses were performed.
Time Frame: Baseline to Week 100
Population: Results are presented for the full analysis set (FAS). FAS included all patients who received at least one dose of study drug in the study eye, had baseline Best Corrected Visual Acuity (BCVA) assessment on the study eye, and had at least one post-baseline BCVA assessment on the study eye.
Measure: Mean (Standard Deviation); unit: letters correctly read
Arm/Group | Open Label IAI
Number analyzed (Participants) | 151
letters correctly read
  Week 100 | 58.7 (20.5)
  Change from Baseline at Week 100 | 4.5 (17.2)

2. Secondary Outcome: Percentage of Participants Whose Optical Coherence Tomography (OCT) Status Was "Dry" at Week 52 and at Week 100 (LOCF)
Description: Retinal fluid status was evaluated using spectral domain OCT on the study eye at every study visit. Last observation carried forward (LOCF) method was used to impute missing data.
Time Frame: Baseline to Week 100
Population: Full analysis set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Open Label IAI
Number analyzed (Participants) | 151
percentage of participants
  Baseline: Dry | 0.7
  Baseline: Not Dry | 99.3
  Week 52: Dry | 53.0
  Week 52: Not Dry | 47.0
  Week 100: Dry | 51.7
  Week 100: Not Dry | 48.3

3. Secondary Outcome: Percentage of Participants Who Gained ≥15 ETDRS Letters Compared With Baseline at Week 52 and Week 100 (LOCF)
Description: as for outcome 1
Time Frame: At week 52 and At week 100
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Open Label IAI
Number analyzed (Participants) | 151
percentage of participants
  At week 52 | 25.8
  At week 100 | 22.5

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity Score Through Week 52 (LOCF)
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision.
Time Frame: Baseline to Week 52
Population: FAS
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Open Label IAI
Number analyzed (Participants) | 151
Letters correctly read
  At Week 52 | 60.1 (18.94)
  Change from Baseline at Week 52 | 5.9 (15.54)

5. Secondary Outcome: Percentage of Participants Who Gained ≥0, ≥5, ≥10, or ≥30 Letters From Baseline in BCVA Through Week 100 (LOCF)
Description: Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better functioning.
Time Frame: Baseline to Week 100
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Open Label IAI
Number analyzed (Participants) | 151
percentage of participants
  Gained ≥ 0 Letters at Week 100 | 70.9
  Gained ≥ 5 Letters at Week 100 | 57.6
  Gained ≥10 Letters at Week 100 | 40.4
  Gained ≥30 Letters at Week 100 | 4.6

6. Secondary Outcome: Percentage of Patients Who Lost >0, ≥5, ≥10, or ≥15 Letters From Baseline in BCVA Through Week 100 (LOCF)
Description: as for outcome 5
Time Frame: Baseline to Week 100
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Open Label IAI
Number analyzed (Participants) | 151
percentage of participants
  Lost >0 Letters at Week 100 | 29.1
  Lost ≥5 Letters at Week 100 | 23.2
  Lost ≥10 Letters at Week 100 | 16.6
  Lost ≥15 Letters at Week 100 | 13.2

7. Other Pre Specified Outcome: Percent Change From Baseline in Corneal Endothelial Cell Density (ECD) at Week 24 and Week 52 in the Study Eye and the Fellow Eye - Endothelial Cell Density Evaluable Set (EES)
Description: EES included all eligible patients who were treated in the study eye, untreated in the fellow eye, had baseline specular microscopy image in both eyes, and completed week 52 evaluation in both eyes and treatment with systemic anti-VEGF therapeutics
Time Frame: At week 24 and At week 52
Population: EES
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Open Label IAI
Number analyzed (Participants) | 118
percent change from baseline
  Week 24: Study eye: number analyzed (Participants) | 106
  Week 24: Study eye | -0.3 (4.15)
  Week 24: Fellow eye: number analyzed (Participants) | 106
  Week 24: Fellow eye | 1.0 (4.28)
  Week 52: Study eye | -0.2 (4.19)
  Week 52: Fellow eye | -0.3 (4.04)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period baseline to week 100
Arm/Group | Open Label IAI
Serious Adverse Events (participants affected / at risk) | 45/154
Other Adverse Events (participants affected / at risk) | 38/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label IAI (N=154)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Thromboangiitis obliterans (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1 — Study eye
Detachment of retinal pigment epithelium (Eye disorders) | 1 — Study eye
Retinal haemorrhage (Eye disorders) | 1 — Study eye
Retinal pigment epithelial tear (Eye disorders) | 1 — Study eye
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 4
Coronary artery disease (Cardiac disorders) | 3
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Endophthalmitis (Infections and infestations) | 1
Endophthalmitis (Infections and infestations) | 1 — Study eye
Gastroenteritis bacterial (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label IAI (N=154)
Hypertension (Vascular disorders) | 13
Conjunctival haemorrhage (Eye disorders) | 12 — Study eye
Neovascular age-related macular degeneration (Eye disorders) | 20
Vitreous detachment (Eye disorders) | 9 — Study eye
Vitreous floaters (Eye disorders) | 9 — Study eye
Bronchitis (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the trial, the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review; provided that the sponsor can remove confidential or proprietary information from such communications. The sponsor cannot require other changes to the communication and cannot extend the embargo.